CLINICAL TRIAL: NCT06454916
Title: GI Windows Flexagon Self Forming Magnet Anastomosis Plus OTOLoc for Creating Small Bowel Anastomoses in Patients Undergoing Surgical Procedures
Brief Title: Functional Lumen Opening With Self-Forming Magnetic Anastomosis
Acronym: FLOWS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GI Windows, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIW 24-001
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Small Bowel Anastomosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Study Group: Prospective Evaluation of the Flexagon SFM Device with OTOLoc (Experimental): This is a multicenter, single-arm study in which clinical outcomes are prospectively evaluated for a minimum of 70 subjects undergoing small bowel anastomosis using the Flexagon SFM Device with OTOLoc.
  Interventions: Device: Small Bowel Anastomosis with Flexagon SFM Device with OTOLoc

INTERVENTIONS:
Device: Small Bowel Anastomosis with Flexagon SFM Device with OTOLoc — This study will investigate one type of intervention: small bowel anastomosis creation in subjects undergoing laparoscopic small bowel surgery. Flexagon SFMs and OTOLoc devices will be delivered laparoscopically into two different sections of small bowel that are intended to be anastomosed. An OTOLoc device will be deployed into the small bowel wall in one section of the small bowel to provide access for the deployment of a Flexagon SFM into that section of bowel. The process is repeated at the second section of bowel. Once deployed, the Flexagon SFMs are approximated and positioned, after which the SFMs are couple together to form the anastomosis, with the OTOLoc devices allowing fluidic communication between the two sections of bowel until the anastomosis is fully formed.

SUMMARY:
The primary objective of this trial is to investigate the safety and effectiveness of the Flexagon SFM system plus OTOLoc when used to create a small bowel anastomosis in subjects undergoing laparoscopic small bowel surgery.

DETAILED DESCRIPTION:
This is a multicenter, pivotal study in which clinical outcomes will be prospectively evaluated for a minimum of 70 subjects undergoing anastomosis creation using the Flexagon SFM system plus OTOLoc.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 22 years or older at screening
2. Candidate for laparoscopic small bowel surgery requiring small bowel anastomosis with cardiac/medical clearance for surgery
3. Able to understand and sign informed consent document
4. American Society of Anesthesiologists (ASA) score < IV at time of procedure
5. Lives, and intends to remain, within a 185-mile radius of study center for the duration of the study
6. Able to refrain from smoking during study follow-up period

Exclusion Criteria:

1. Known or suspected allergy to silicone, nickel, titanium or Nitinol
2. BMI > 55 kg/m2
3. Uncontrolled diabetes (defined as HbA1c >10%)
4. Congenital or acquired anomalies of the GI tract, including atresia or malrotation
5. Diagnosed with obstructed or perforated colon cancer
6. Any documented conditions for which endoscopy and/or laparoscopy would be contraindicated or history of previous technically difficult or failed endoscopy
7. Any previous major surgery on the stomach, duodenum, hepatobiliary tree (excluding laparoscopically removed gallbladder or prior sleeve gastrectomy), pancreas or right colon
8. Coagulation deficiency not normalized by medical treatment or platelet count <50,000/µL
9. Known moderate to severe renal disease (eGFR < 44 milliliters per minute per 1.73m2) or ongoing dialysis
10. Hyperkalemia / hypercoagulability or prior Venus Thromboembolism / Pulmonary Embolism
11. Immunocompromised (e.g., active treatment for malignancies, hematologic malignancy, on immunosuppressive therapy, moderate or severe primary immunodeficiency, advanced or untreated HIV, active treatment with high-dose corticosteroids (i.e., 20 or more mg of prednisone or equivalent per day when administered for 2 or more weeks prior to surgery) or other immunosuppressive or immunomodulatory agents
12. Active H. pylori infection
13. Active or suspected infection at the surgical site or a CDC Class 3/contaminated or Class 4/dirty-infected surgical wound.
14. Obstructive Sleep Apnea on CPAP unless assessed and cleared by independent physician
15. Contraindication to general anesthesia
16. Breast-feeding, pregnant, or planning on becoming pregnant during the follow-up period
17. Currently participating or has participated in another clinical trial within the past 30 days and is receiving/has received an investigational drug, device, or biologic agent
18. Subject is not appropriate for inclusion in the clinical trial, per the medical opinion of the Principal Investigator

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Successful Anastomosis Creation without the Need for Reoperation | 30 Days
  The study's primary endpoint (patient success) is defined as successful anastomosis created with the Flexagon SFM without placement procedure, device or target anastomosis-related reoperation through 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Wilson, MD, Study Chair — The University of Texas Health Science Center, Houston
Locations (7):
- United States (7):
  - Fresno Community Hospital and Medical Center, Clovis, California
  - University of Miami, Coral Gables, Florida
  - Orlando Health, Orlando, Florida
  - Endeavor Health, Evanston, Illinois
  - Duke Regional Hospital, Durham, North Carolina
  - UT Health Houston, Houston, Texas
  - Seger Bariatrics and Metabolism, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.